CLINICAL TRIAL: NCT05988346
Title: Ghrelin Expression Could Regulate Diastolic Heart Function in Obese Patients With Diabetes
Brief Title: Ghrelin and Diastolic Heart Function
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, Professor of Medicine, University of Campania Luigi Vanvitelli
Other Study IDs: 0408052023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2; Obesity, Abdominal; Diastolic Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Authors will analyze biospecimen from the removed abdominal adipose tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- type 2 diabetes mellitus (T2DM) obese patients without left ventricle (LV) diastolic dysfunction.
  Interventions: Procedure: abdominal plastic intervention
- T2DM obese patients with first degree of left ventricle (LV) diastolic dysfunction.
  Interventions: Procedure: abdominal plastic intervention
- T2DM obese patients with second degree of left ventricle (LV) diastolic dysfunction.
  Interventions: Procedure: abdominal plastic intervention

INTERVENTIONS:
Procedure: abdominal plastic intervention — According to international guidelines, authors will remove the superficial abdominal fat from the patients enrolled in the study.

SUMMARY:
In type 2 diabetes mellitus (T2DM) and obese patients the adipose tissue could over-express cytokines, sirtuin-1 (SIRT1), and microRNAs (miRs) implied in the regulation of left ventricle (LV) diastolic function (LV-DF). Ghrelin could modulate these pathways. Thus, in the current study authors will investigate ghrelin expression in T2DM obese patients after abdominal fat excision, and particularly in those with normalization of LV-DF at 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM obese patients;
* T2DM obese patients under anti-diabetic full medical therapy and glycemic control.

Exclusion Criteria:

* clinical diagnosis of type 1 diabetes;
* T2DM patients in poor glycemic control (HbA1c values of >7%);
* chronic neurological disorders;
* heart failure and coronary heart disease or depression of left ventricular ejection fraction (LVEF <55%);
* severe anemia;
* thyroid dysfunction;
* kidney failure;
* uncontrolled blood pressure (blood pressure > 140/90 mmHg on two occasions 2 weeks apart);
* inflammatory chronic disease;
* neoplastic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The authors will enroll T2DM obese patients, according to the evidence or not of LV diastolic dysfunction, and then divided in three groups. The LV diastolic dysfunction was characterized as indicated by international recommendations, by the values of E/E' ratio (18). Thus, the patients without LV diastolic dysfunction (E/E'<9) were characterized as group 1. Those with LV diastolic dysfunction (E/E'>9), were divided in two groups, in accordance with the E/E' values: group 2 (the patients with 9<E/E'<13), and group 3 (the patients with E/E'>13).
  Obesity will be diagnosed as body mass index (BMI) > 30 (15). All enrolled patients will have T2DM according to international guidelines diagnostic criteria: evidence of fasting plasma glucose of ≥7.0 mmol/L (126 mg/dL; impaired fasting glucose [IFG]), a 2-hour glucose of ≥11.1 mmol/L during a 75 g oral glucose tolerance test (GTT) (>200 mg/dL; impaired glucose tolerance [IGT]), or a plasma hemoglobin (Hb) A1c of ≥48 mmol/mol (≥6.5%), (16).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
normalization of LV diastolic dysfunction | 12 months
  At 1 year of follow-up authors evaluated the patients (those with first and second degree of LV diastolic dysfunction) that will experience the normalization of LV diastolic function.

CONTACTS AND LOCATIONS:
Locations (1):
- Celestino Sardu, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, D'Onofrio N, Trotta MC, Balestrieri ML, Nicoletti GF, D'Amico G, Fumagalli C, Contaldi C, Pacileo G, Scisciola L, Nicoletti M, Marfella LV, Sbriscia M, Sasso FC, Signoriello G, Paolisso G, Marfella R. Could Ghrelin Expression Regulate Diastolic Cardiac Function in Type 2 Diabetic Obese Patients? Diabetes Metab Res Rev. 2025 May;41(4):e70049. doi: 10.1002/dmrr.70049. PMID 40323144